CLINICAL TRIAL: NCT03637205
Title: Prospective Randomized Multicenter Study Comparing Extracorporeal Life Support Plus Optimal Medical Care Versus Optimal Medical Care Alone in Patients With Acute Myocardial Infarction Complicated by Cardiogenic Shock Undergoing Revascularization
Brief Title: Extracorporeal Life Support in Cardiogenic Shock
Acronym: ECLS-SHOCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Health Institute GmbH (Other)
Collaborators: Heart Center Leipzig - University Hospital (Other); IHF GmbH - Institut für Herzinfarktforschung (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRC[045584]
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Acute Myocardial Infarction; Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECLS (Experimental): PCI (or CABG) plus medical treatment + ECLS
  Interventions: Procedure: ECLS insertion; Other: Revascularisation and optimal medical treatment
- No ECLS (Active Comparator): PCI (or CABG) plus medical treatment
  Interventions: Other: Revascularisation and optimal medical treatment

INTERVENTIONS:
Procedure: ECLS insertion — After diagnostic angiography the culprit lesion should be identified and revascularization (preferably by PCI, alternatively CABG) should be planned. ECLS insertion should be performed preferably before revascularization
  Arms: ECLS
Other: Revascularisation and optimal medical treatment — After diagnostic angiography the culprit lesion should be identified and revascularization (preferably by PCI, alternatively CABG) should be planned.

SUMMARY:
The aim of the study is to examine whether treatment with extracorporeal life support (ECLS) in addition to revascularization with percutaneous coronary intervention (PCI) or alternatively coronary artery bypass grafting (CABG) and optimal medical treatment is beneficial in comparison to no ECLS in patients with severe infarctrelated cardiogenic shock with respect to 30-day mortality

ELIGIBILITY:
Inclusion Criteria:

* Cardiogenic shock complicating AMI (STEMI or NSTEMI) plus obligatory:
* Planned revascularization (PCI or alternatively CABG)
* Systolic blood pressure <90 mmHg >30 min or catecholamines required to maintain pressure >90 mmHg during Systole
* Signs of impaired organ perfusion with at least one of the following criteria a) Altered mental Status, b) Cold, clammy skin and extremities, c) Oliguria with urine output <30 ml/h
* Arterial lactate >3 mmol/l
* Informed consent

Exclusion Criteria:

* Resuscitation >45 minutes
* Mechanical cause of cardiogenic shock
* Onset of shock >12 h
* Severe peripheral artery disease with impossibility to insert ECLS cannulae
* Age <18 years or age >75 years
* Shock of other cause (bradycardia, sepsis, hypovolemia, etc.)
* Other severe concomitant disease with limited life expectancy <6 months
* Pregnancy
* Participation in another trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  30-day all-cause death after randomization according to the intention-to-treat principle

SECONDARY OUTCOMES:
Time to death within 6 and 12 months follow-up | 6 and 12 months
Length of mechanical ventilation | 0 to 10 days
Time to hemodynamic stabilization | 0 to 10 days
Duration of catecholamine therapy | 0 to 10 days
Serial creatinine-level and creatinine-clearance | 0 to 10 days from time of randomization until stabilization
  Creatinine-clearance (Cockcroft-Gault-Formula)
Length of ICU stay | 0 to 11 days
Length of hospital stay | 0 to 14 days
Serial SAPS-II score | 0 to 11 days
Mean and area under the curve of arterial lactate | 0 to 14 days
Acute renal failure requiring renal replacement therapy | 0 to 14 days
Cerebral performance category (CPC) | 30 days, 6 and 12 months
Cardiovascular mortality | 6 and 12 months
Hospitalization for heart failure | 6 and 12 months
Recurrent infarction | 30 days, 6 and 12 months
Repeat revascularization (PCI or CABG) | 30 days, 6 and 12 months
Status of Quality of life measured by EQ-5D-5L descriptive system | 12 months
  The EQ-5D-5L descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems expressed by 1-digit-numbers ranging from 1 (extreme problems) to 5 (no problems). The toal score ranges from 0-15 where 15 is the worst score.
Status of Quality of life measured by EQ VAS | 12 months
  The EuroQol Group visual analogue scale (EQ VAS) records the patient's self-rated health on a vertical visual analogue scale from 0 to 100, where the maximum 100 is labelled 'The best health you can imagine' and the minimum 0 is labelled 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, MD, Principal Investigator — Director, Department of Cardiology, Heart Center Leipzig
Locations (46):
- Germany (45):
  - Universitätsklinikum Aachen, Aachen
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - SLK-Kliniken Heilbronn GmbH Klinikum Am Plattenwald, Bad Friedrichshall
  - Kerckhoff-Klinik Forschungsgesellschaft mbH, Bad Nauheim
  - Charité Universitätsmedizin Berlin, CBF Medizinische Klinik für Kardiologie, Berlin
  - BG Klinikum Unfallkrankenhaus Berlin gGmbH, Berlin
  - Universitätsklinikum Köln Klinik III für Innere Medizin, Cologne
  - St-Johannes-Hospital Klinik für Innere Medizin I, Dortmund
  - Technische Universität Dresden, Dresden
  - Universitätsklinikum Düsseldorf Klinik für Kardiologie, Pneumologie und Angiologie, Düsseldorf
  - Helios Klinikum Erfurt 3. Medizinische Klinik, Erfurt
  - Elisabeth-Krankenhaus GmbH Klinik für Kardiologie und Angiologie, Essen
  - Universitätsklinikum Essen (AöR) Westdeutsches Herz- und Gefäßzentrum Essen, Essen
  - Universitätsklinikum Frankfurt ZIM - Med. Klink III - Kardiologie, Frankfurt
  - Klinikum Frankfurt Höchst, Frankfurt Höchst
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen und Innere Medizin III - internistische Intensivmedizin, Freiburg im Breisgau
  - Universitätsklinikum Gießen, Giessen
  - Universitätsmedizin Göttingen Klinik für Kardiologie und Pneumologie, Göttingen
  - Universitätsmedizin Greifswald, Greifswald
  - Universitätsklinikum Halle (Saale) Universitätsklinik und Poliklinik für Innere Medizin III, Halle
  - Asklepios Kliniken Hamburg GmbH, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf Klinik für Kardiologie, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Universitätsklinikum des Saarlandes Klinik für Innere Medizin III, Homburg
  - Uniklinikum Jena Klinik für Innere Medizin I, Jena
  - Klinikum Kassel GmbH, Kassel
  - Helios Klinikum Krefeld, Krefeld
  - Asklepios Kliniken Langen-Seligenstadt GmbH, Langen
  - Universität Leipzig Klinik und Poliklinik für Kardiologie, Leipzig
  - Herzzentrum Leipzig, Leipzig
  - Klinikum der Stadt Ludwigshafen gGmbH, Ludwigshafen
  - Universitäres Herzzentrum Lübeck Medizinische Klinik II (Kardiologie, Angiologie, Intensivmedizin), Lübeck
  - Universitätsmedizin Mannheim, Mannheim
  - Kliniken Mariahilf GmbH, Mönchengladbach
  - Klinikum Nürnberg, Nuremberg
  - Universitätsklinikum Regensburg Klinik und Poliklinik für Innere Medizin II, Regensburg
  - Kreiskliniken Reutlingen GmbH, Reutlingen
  - Universitätsmedizin Rostock Zentrum für Innere Medizin, Rostock
  - Helios Klinikum Siegburg, Siegburg
  - Universitätsklinikum Ulm Klinik für Innere Medizin II / Kardiologie, Ulm
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden GmbH Klinik Innere MED I: Kardiologie und konserv. Intensivmedizin, Wiesbaden
  - Rems-Murr-Kliniken Winnenden Abteilung für Kardiologie, Winnenden
  - Helios Universitätsklinikum Wuppertal Medizinische Klinik 3 - Kardiologie, Wuppertal
  - Universitätsklinikum Würzburg Medizinische Klinik und Poliklinik I, Würzburg
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thevathasan T, Alyahoud M, Freund A, Akin I, Fichtlscherer S, Zeymer U, Feistritzer HJ, Poss J, Jobs A, Rossberg M, Jung C, Skurk C, Rassaf T, Ouarrak T, Schneider S, Thiele H, Desch S. Extracorporeal Membrane Oxygenation Complications Are Not Causal for Mortality in Patients With Infarct-Related Cardiogenic Shock: A Mediation Analysis of the Extracorporeal Life Support in Infarct-Related Cardiogenic Shock (ECLS-SHOCK) Trial. Crit Care Med. 2025 Dec 1;53(12):e2607-e2617. doi: 10.1097/CCM.0000000000006893. Epub 2025 Oct 17. PMID 41114622
- [Derived] Feistritzer HJ, Zeymer U, Ouarrak T, Akin I, Rassaf T, Lehmann R, Eitel I, Seidler T, Skurk C, Clemmensen P, Voigt I, Seyfarth M, Linke A, Tigges E, Jung C, Lauten P, Poss J, Schneider S, Desch S, Freund A, Thiele H; ECLS-SHOCK Investigators. Different Mechanical Circulatory Support Strategies for Infarct-Related Cardiogenic Shock: A Subanalysis of the ECLS-SHOCK Trial. JACC Cardiovasc Interv. 2025 Mar 24;18(6):691-701. doi: 10.1016/j.jcin.2024.12.010. PMID 40139846
- [Derived] Thiele H, Zeymer U, Akin I, Behnes M, Rassaf T, Mahabadi AA, Lehmann R, Eitel I, Graf T, Seidler T, Schuster A, Skurk C, Duerschmied D, Clemmensen P, Hennersdorf M, Fichtlscherer S, Voigt I, Seyfarth M, John S, Ewen S, Linke A, Tigges E, Nordbeck P, Bruch L, Jung C, Franz J, Lauten P, Goslar T, Feistritzer HJ, Poss J, Kirchhof E, Ouarrak T, Schneider S, Desch S, Freund A; ECLS-SHOCK Investigators. Extracorporeal Life Support in Infarct-Related Cardiogenic Shock. N Engl J Med. 2023 Oct 5;389(14):1286-1297. doi: 10.1056/NEJMoa2307227. Epub 2023 Aug 26. PMID 37634145